CLINICAL TRIAL: NCT04494438
Title: Rituximab in Patients With Low Dose Steroid-dependent Idiopathic Nephrotic Syndrome
Brief Title: Rituximab for Idiopathic Nephrotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, Principal Investigator, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGG-SN-MAB2 Low Dose
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Idiopathic Nephrotic Syndrome
Keywords: Nephrotic syndrome; Proteinuria; Rituximab
MeSH Terms: conditions — Nephrosis, Lipoid; Nephrotic Syndrome; Proteinuria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid tapering. (No Intervention)
- Rituximab (Experimental): Single administration of Rituximab 375 mg/mq at a rate of 0.5 to 1.5 ml/min over approximately 6 hours, following the infusion of 2.5-5 mg of intravenous chlorfenamine maleate (based on the local protocol and patient tolerance), methylprednisolone (2 mg/Kg) in normal saline and oral paracetamol (8 mg/kg).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: Mabthera; Anti CD-20 antibodies
  Arms: Rituximab

SUMMARY:
Open-label, randomized, controlled trial due to value whether the monoclonal antibody rituximab is non-inferior to steroids in maintaining remission in juvenile forms of SDNS.

The investigators will enroll 30 pediatric patients affected by idiopathic nephrotic syndrome, who have been in treatment with steroids for at least one year. The lowest dose of drug required to maintain a stable remission will be between 0.4 and 0.7 mg/ kg/ day.

This trial provides an initial run-in phase of one month during wich remission will be achieved by means of a standard oral prednisone course. Once remission has been achieved children will be randomized in a parallel arm open label RCT to continue prednisone alone for one month (control) or to add a single intravenous infusion of rituximab (375 mg/m2 - intervention). Prednisone will be tapered in both arms after one month.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 16 years.
* Steroid-dependent idiopatic nephrotic syndrome for a minimum of 6 to a maximum of 12 months at the time of study entry, regardless of disease duration.
* Low-dose steroid dependence (between 0.4 and 0.7 mg/ kg/ day)

Exclusion Criteria:

* Positivity of autoimmunity tests (ANA, nDNA, ANCA) or reduced C3 levels
* Histological pattern suggestive for congenital anomalies (diffuse mesangial sclerosis without IgM deposits, cystic-like tubular dilations, evidence of mithocondrial damage on electronic microscopy.
* Histological pattern not correlated with idiopathic nephrotic syndrome in the pediatric age (membranous glomerulonephritis, lupus nephritis, diffuse and/or localized vasculitis, amyloidosis).
* Evidence of homozygous or heterozygous mutations in podocitary genes commonly involved in the pathology (NPHS1, NPHS2, WT1).
* Estimated glomerula filtration rate (eGFR) < 60ml/min.
* Presence of circulating IgM against HCV, HBV, parvovirus or mycoplasm.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Three months proteinuria | 3 months
  To be considered non-inferior, rituximab will have to allow steroid withdrawal and maintain three-month proteinuria within a pre-specified non-inferiority margin of three times the levels among controls.

SECONDARY OUTCOMES:
Time-to-relapse mesaure | 12 months
  Risk of relapse of proteinuria and need for recovery of steroids, with survival analysis after withdrawal of steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco Ghiggeri, MD, Study Director — Istituto Giannina Gaslini
Locations (1):
- IRCCS Giannina Gaslini Institute, Genova, Italy

REFERENCES:
- [Background] Ravani P, Ponticelli A, Siciliano C, Fornoni A, Magnasco A, Sica F, Bodria M, Caridi G, Wei C, Belingheri M, Ghio L, Merscher-Gomez S, Edefonti A, Pasini A, Montini G, Murtas C, Wang X, Muruve D, Vaglio A, Martorana D, Pani A, Scolari F, Reiser J, Ghiggeri GM. Rituximab is a safe and effective long-term treatment for children with steroid and calcineurin inhibitor-dependent idiopathic nephrotic syndrome. Kidney Int. 2013 Nov;84(5):1025-33. doi: 10.1038/ki.2013.211. Epub 2013 Jun 5. PMID 23739238
- [Background] Ghiggeri GM, Musante L, Candiano G, Bruschi M, Santucci L, Barbano G, Trivelli A, Rivabella L, Gusmano R, Perfumo F. Protracted remission of proteinuria after combined therapy with plasmapheresis and anti-CD20 antibodies/cyclophosphamide in a child with oligoclonal IgM and glomerulosclerosis. Pediatr Nephrol. 2007 Nov;22(11):1953-6. doi: 10.1007/s00467-007-0550-y. Epub 2007 Jul 28. PMID 17661091
- [Background] Pescovitz MD, Book BK, Sidner RA. Resolution of recurrent focal segmental glomerulosclerosis proteinuria after rituximab treatment. N Engl J Med. 2006 May 4;354(18):1961-3. doi: 10.1056/NEJMc055495. No abstract available. PMID 16672715
- [Background] Magnasco A, Ravani P, Edefonti A, Murer L, Ghio L, Belingheri M, Benetti E, Murtas C, Messina G, Massella L, Porcellini MG, Montagna M, Regazzi M, Scolari F, Ghiggeri GM. Rituximab in children with resistant idiopathic nephrotic syndrome. J Am Soc Nephrol. 2012 Jun;23(6):1117-24. doi: 10.1681/ASN.2011080775. Epub 2012 May 10. PMID 22581994
- [Background] Ravani P, Magnasco A, Edefonti A, Murer L, Rossi R, Ghio L, Benetti E, Scozzola F, Pasini A, Dallera N, Sica F, Belingheri M, Scolari F, Ghiggeri GM. Short-term effects of rituximab in children with steroid- and calcineurin-dependent nephrotic syndrome: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1308-15. doi: 10.2215/CJN.09421010. Epub 2011 May 12. PMID 21566104
- [Background] Ruggenenti P, Ruggiero B, Cravedi P, Vivarelli M, Massella L, Marasa M, Chianca A, Rubis N, Ene-Iordache B, Rudnicki M, Pollastro RM, Capasso G, Pisani A, Pennesi M, Emma F, Remuzzi G; Rituximab in Nephrotic Syndrome of Steroid-Dependent or Frequently Relapsing Minimal Change Disease Or Focal Segmental Glomerulosclerosis (NEMO) Study Group. Rituximab in steroid-dependent or frequently relapsing idiopathic nephrotic syndrome. J Am Soc Nephrol. 2014 Apr;25(4):850-63. doi: 10.1681/ASN.2013030251. Epub 2014 Jan 30. PMID 24480824
- [Background] Guigonis V, Dallocchio A, Baudouin V, Dehennault M, Hachon-Le Camus C, Afanetti M, Groothoff J, Llanas B, Niaudet P, Nivet H, Raynaud N, Taque S, Ronco P, Bouissou F. Rituximab treatment for severe steroid- or cyclosporine-dependent nephrotic syndrome: a multicentric series of 22 cases. Pediatr Nephrol. 2008 Aug;23(8):1269-79. doi: 10.1007/s00467-008-0814-1. Epub 2008 May 9. PMID 18465150
- [Background] Fernandez-Fresnedo G, Segarra A, Gonzalez E, Alexandru S, Delgado R, Ramos N, Egido J, Praga M; Trabajo de Enfermedades Glomerulares de la Sociedad Espanola de Nefrologia (GLOSEN). Rituximab treatment of adult patients with steroid-resistant focal segmental glomerulosclerosis. Clin J Am Soc Nephrol. 2009 Aug;4(8):1317-23. doi: 10.2215/CJN.00570109. Epub 2009 Jul 2. PMID 19578004
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526